CLINICAL TRIAL: NCT05865548
Title: Randomized Control Trial of Addition of Aspirin to Standard Care in Oral Cancer Patients.
Brief Title: Addition of Aspirin to Standard of Care in Oral Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Banaras Hindu University (Other)
Responsible Party: Principal Investigator, Manoj Pandey, Professor, Banaras Hindu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNC02
Record Dates: First submitted 2023-04-28; First posted 2023-05-19 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms | interventions — Aspirin; Standard of Care; Radiation; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Two arm study comparing standard of care with or without aspirin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Experimental): Aspirin 150mg PO daily along with standard of care
  Interventions: Drug: Aspirin 150 mg
- Standard of care (Active Comparator): Standard of care as per the stage of disease and guidelines i.e. Surgery, Surgery with radiation or palliative chemotherapy as per investigators choice
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Drug: Aspirin 150 mg — Aspirin 150 mg PO daily
  Arms: Interventional arm
Procedure: Standard of care — Surgery with or without radiation, palliative chemo as per investigators choice
  Other Names: Radiation, chemotherapy
  Arms: Standard of care

SUMMARY:
Despite accumulating evidence of the benefit of aspirin in cancer, its effect on improving cancer survival is still debated since the mechanism by which it impacts cancer survival is not completely understood and the published data are discordant. There have been 4 randomized controlled trials (RCT) showing mixed results from no effect to improved survival. Several retrospective and observational studies have reported a survival advantage of adding aspirin to the treatment for various cancers. A meta-analysis of 118 studies, 63 of them specifically reporting on cancer mortality and the rest on all-cause mortality, found a 21% reduction in cancer deaths and about 20% reduction in all-cause mortality (pooled hazard ratio (HR): 0.79; 95% confidence intervals: 0.73, 0.84).

However, the evidence is still lacking and there is need to do more RCT

DETAILED DESCRIPTION:
Aspirin (ASA), an NSAID, is a well-known antipyretic and analgesic agent and is used to prevent recurrent transient ischemic attacks or strokes. In addition to its classical anti- inflammatory function, clinical and epidemiological studies indicate that aspirin can be used as a preventive or therapeutic agent in multiple cancers, including oral cancers

While the exact mechanism through which NSAIDs contribute to chemo prevention is not completely understood, Aspirin inhibits the enzyme Cox; Cox-1 and Cox-2 are well characterized. Cox converts a arachidonic acid to prostaglandin H2, which in turn produces biologically active prostaglandins that influence path physiological processes in a range of tissues including angiogenesis, apoptosis, cell proliferation and migration, inflammatory response and thrombosis. Inhibition of prostaglandin synthesis is considered the pre dominant mechanism by which NSAIDs act as anti-inflammatory agents, but it is unclear whether the anti-cancer properties of these agents can be solely attributed to Cox inhibition.

Recently, Cox-2 over expression has been identified in a number of different malignancies and it has been hypothesized that Cox-2 prostaglandins promote tumor genesis by inhibiting apoptosis, modulating the immune system and regulating tumor associated angiogenesis.

A detailed search of literature and bio informatics analysis of the data obtained showed that the effect of Aspirin on survival and prevention of recurrence and secondary cancer could be due to its effect on following 11 genes PTGS2, PIK3CA, PARP1, PARP2, VEGFA, KDR, PTGES2, NFKB1, P53, FLT1, VEGFR. These genes not only interact and control each other but also control cell cycle regulation through other genes as shown below. These could be due to co expression, physical interactions, shared domains or predicted interactions in absence of data.

Based on the gene-gene and protein-protein interactions they can be clustered into three with PTGES2, PTGS2 and p53 being in first cluster (figure 2 below), the NGS data obtained from the previous patients also showed the p53 to be the primary driver gene (unpublished data, submitted) in nearly 50% of the subjects. It has also been shown that patients with p53 mutations

have poor survival and increased recurrence rates compared to those without p53 mutations. This coupled with literature showing improved survival and low recurrence in patients receiving Aspirin suggest the need for a RCT as this has never been done before.

ELIGIBILITY:
Inclusion Criteria:

* All Histologically proven cases of primary oral cancers.
* Stage T1 to T4, N0 to N3, M0 to M1.
* Age above 18.
* Karnofsky' performance status more than 70, ECOG 0 to 2
* Hb >8.0 gm/dL
* Total count >4000 cu mm
* Platelet count >100000 Serum creatinine <1.0mg
* Liver enzymes up to 1.5 times normal
* Bilirubin <1.0mg

Exclusion Criteria:

* Patients with acid peptic disease
* Pregnant and lactating women.
* Patients not willing to participate.
* Patients with known allergy to NSAID
* Patients with Asthma, rhinitis and nasal polyps
* Presence of viral fever
* Use of any other blood thinner like warfarin, heparin or low molecular weight heparin
* bleeding/blood-clotting disorders (such as hemophilia, vitamin K deficiency, low platelet count)
* pyruvate kinase or G6PD deficiency
* Patients receiving mifepristone, acetazolamide, corticosteroids, dichlorphenamide, methotrexate, valproic acid, herbal medications (such as ginkgo biloba)
* Patients with recent history of anti-viral vaccines

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Adverse events | 4 weeks
  Number of participants with treatment-related adverse events as assessed by WHO toxicity criteria

SECONDARY OUTCOMES:
Disease free survival | through study completion, an average of 2 year
  Local recurrence or metastasis from the time from the diagnosis to the closer of study
Overall survival | through study completion, an average of 2 year
  Death from the time of diagnosis to closer of study

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Pandey, Principal Investigator — Professor
Locations (1):
- Banaras Hindu University, Varanasi, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No